CLINICAL TRIAL: NCT01547442
Title: Artisan Aphakia Lens for the Correction of Aphakia in Children
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Ophtec USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Artisan Pediatric Aphakia
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Aphakia
Keywords: aphakia; secondary intraocular lens; congenital cataract; marfan syndrome; pediatric cataract; ectopia lentis; subluxated lens
MeSH Terms: conditions — Aphakia; Marfan Syndrome; Ectopia Lentis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artisan Aphakia Intraocular Lens (Experimental): Implantation of an Artisan intraocular lens to correct aphakia in children
  Interventions: Device: Artisan Aphakia Intraocular Lens

INTERVENTIONS:
Device: Artisan Aphakia Intraocular Lens — Implantation of an intraocular lens

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Artisan Aphakia Lens in the treatment of aphakia in children.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 21 years of age
* Have a visually significant cataract or need IOL replacement surgery
* Compromised capsular bag prohibiting implantation of standard posterior IOL
* Subject or parent/guardian must be able to comply with visit schedule and study requirements
* Subject's legal representative must be able to sign the Informed Consent

Exclusion Criteria:

* Under 2 years of age
* Unable to meet Postoperative evaluation requirements
* No useful vision or vision potential in fellow eye
* Mentally retarded patients
* History of corneal disease
* Abnormality of the iris or ocular structure
* ACD less than 3.2 mm
* Uncontrolled glaucoma
* IOP > 25 mmHg
* Chronic or recurrent uveitis
* Preexisting macular pathology that may complicate the ability to assess the benefit of this lens
* Retinal detachment or family history
* Retinal disease that may limit visual potential
* Optic nerve disease that may limit visual potential
* Diabetes mellitus
* Pregnant, lactating or plan to become pregnant

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected distance visual acuity at 12 months postoperative | 5 years follow up
  Determination of the ability of the lens to correct refractive error caused by aphakia

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Farhan, Study Director — Sponsor GmbH
Locations (19):
- United States (18):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - The Vision Center, Los Angeles, California
  - Indiana University, Riley Hospital for Children, Indianapolis, Indiana
  - Harvard University, Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, MN Lions Children's Eye Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Washington University, St. Louis Children's Hospital, St Louis, Missouri
  - Rosenthal Eye and Facial Plastic Surgery, Great Neck, New York
  - New York Medical College, Westchester Medical Center, Valhalla, New York
  - Nationwide Children's Hospital, Pediatric Ophthalmology Associates, Columbus, Ohio
  - University Hospitals Case Medical Center, Rainbow Babies and Children's Hospital, Mayfield Heights, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - University of Texas, Robert Cizik Eye Clinic, Houston, Texas
  - Moran Eye Center, Salt Lake City, Utah
- Credit Valley Eyecare, Mississauga, Ontario, Canada